CLINICAL TRIAL: NCT04143230
Title: Accuracy of a New Simplified Screening Tool in Identifying the In-hospital Patients in Need of Palliative Care
Brief Title: Identification of In-hospital Patients in Need of Palliative Care Using a New Simplified Screening Tool
Acronym: SST2017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Paolo Cotogni, Head of Acute Palliative Care Unit and Palliative Care Team, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0014892
Record Dates: First submitted 2019-10-15; First posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Locally Advanced Cancer; Metastatic Cancer; Chronic Respiratory Failure; Chronic Heart Failure; Chronic Liver Failure; Chronic Renal Failure
Keywords: palliative care; palliative care team; palliative care unit; screening tool; end of life; unplanned hospital admission; end-stage disease; cancer; survival; prognostic score; palliative sedation
MeSH Terms: conditions — Neoplasm Metastasis; End Stage Liver Disease; Kidney Failure, Chronic; Death; Neoplasms | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: Eligible patients will be evaluated for the need of palliative care, randomly by means of the EST screening tool (ARM A) or by means of the Simplified Screening Tool (SST), (ARM B).
Who Masked: Participant, Care Provider
Masking Description: The Principal Investigator provided close envelops containing the SIAARTI/NCCN screening tool or the Simplified Screening Tool. The screening tool was inserted in the envelop according with a randomization list. The sub-investigator who wold examine the patient had to take the close envelope marked with the corresponding progressive number of patient enrolled, without possibility of choose the tool.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extended Screening Tool (EST) (Active Comparator): The SIAARTI/NCCN (EST) screening tool is, in fact, an instrument validated by many scientific societies, but it is very articulated and its compilation is too much time-consuming.
  Interventions: Other: Screening for PC by means of two different screening tools
- Simplified Screening Tool (SST) (Experimental): The Simplified Screening Tool (SST) has been created through a statistical process in order to include all the critical variables, with the advantage of being shorter and therefore easier to administer in a routinely use.
  Interventions: Other: Screening for PC by means of two different screening tools

INTERVENTIONS:
Other: Screening for PC by means of two different screening tools — Screening of chronically ill patients admitted to an Internal Medicine Unit from the Emergency Department, for palliative care need, using of both the SIAARTI/NCCN screening tool (EST), and the Simplified Screening Tool (SST), derived from the first instrument.

SUMMARY:
Every day many patients affected by chronic life-limiting illnesses are admitted into Internal Medicine wards, coming from the Emergency Department. Many studies suggest that providing palliative care to these patients may improve their end-of-life care while reducing costs by minimizing futile treatments and unwanted intensive care unit admissions. Consequently, there is a strong need for acute care hospitals to more vigorously identify patients entering the final phase of their lives as well as their specific care needs.

In a previous study the investigators screened for need of palliative care patients affected by progressive chronic diseases by means of a tool, based on the Italian Society of Anesthesia, Analgesia, Resuscitation, and Intensive Care - SIAARTI - position paper reporting criteria for patients with end-stage chronic organ failures, and on the specific clinical indicators elaborated by the National Comprehensive Cancer Network (NCCN) for patients with locally advanced/metastatic cancer. In a further pilot study, the investigators compared the outcomes of PC patients depending on whether the palliative care team evaluated such patients only if requested by the physician staff or routinely, irrespectively of a specific request, finding a significant increase of discharges after the activation of an appropriate PC service or scheduled PC ambulatory visit.

In the present study the investigators enroll chronically ill patients admitted to an Internal Medicine Unit from the Emergency Department, to be screened for palliative care need, using the previously cited SIAARTI/NCCN screening tool (Extended Screening Tool - EST), or using a Simplified Screening Tool (SST), derived from the first instrument, which preliminary showed a superimposable efficacy. This latter tool has advantages related to much more shortness and therefore simplicity in the administration to a seriously ill patient and is much less time consuming, allowing the physician to use it routinely.

The aim of the study is to verify the accuracy of the SST in identifying chronically ill patients in need of a PC approach, in comparison to the SIAARTI/NCCN tool (EST). If the SST would show good accuracy, an easily manageable tool for the assessment of PC needs in chronically ill patients would be available for the daily routine.

DETAILED DESCRIPTION:
Due to population aging and advances in medicine and public health, the prevalence of people affected by progressive, chronic, life-limiting diseases is increasing. Many studies documented that patients with progressive chronic diseases received care that was more aimed at the prolongation of life than palliation of symptoms during their last 6-12 months of life, as well as frequent hospitalizations. These data suggested that providing palliative care (PC) to these patients may improve their end-of-life care while reducing costs by minimizing futile treatments and unwanted ICU care.

Consequently, there is a strong need for acute care hospitals to more vigorously identify patients entering the final phase of their lives as well as their specific care needs.

Historically, Hospice and PC services have focused on the needs of cancer patients. However, the majority of patients needing PC worldwide suffer from life-limiting non-cancer illnesses, like cardiovascular diseases, chronic obstructive pulmonary disease (COPD), renal failure, cirrhosis of the liver, Alzheimer's and other dementias, multiple sclerosis, Parkinson's disease, HIV/AIDS, rheumatoid arthritis, and diabetes. The main illnesses requiring PC are cardiovascular diseases (38%), cancer (34%), and COPD (10%).

In order to correctly identify such patients, adequate screening tools are needed.

In a previous study, the investigators employed for this aim a screening tool derived from the Italian Society of Anesthesia, Analgesia, Resuscitation, and Intensive Care (SIAARTI) position paper based on expert panel opinions reporting criteria to identify patients with end-stage chronic organ failures. For cancer patients, the screening was done according to specific clinical indicators elaborated by the National Comprehensive Cancer Network (NCCN). A Simplified Screening Tool was also created, in order to make available an easier instrument for the same aim.

The SIAARTI/NCCN screening tool (Extended Screening Tool - EST) is, in fact, an instrument validated by many scientific societies, but it is very articulated and its compilation is too much time-consuming. The Simplified Screening Tool (SST) has been created through a statistical process in order to include all the critical variables, with the advantage of being shorter and therefore easier to administer in a routinely use.

The aim of the current study is to demonstrate that the SST has accuracy comparable to that of the SIAARTI/NCCN tool in identifying chronically ill patients in need of a PC approach, thus making available an easily manageable tool for the assessment of PC needs in chronically ill patients.

In order to do this, every enrolled patient will be administered both the SST and the SIAARTI/NCCN tool, in a randomized sequence.

After completion of the enrollment and data collection, an appropriate statistical methodology will be employed for the comparison between the established SIAARTI/NCCN tool and the SST.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted to Molinette Hospital (A.O.U. "Città della Salute e della Scienza"), affected by:

* locally advanced/metastatic cancer not suitable to antineoplastic therapy
* locally advanced/metastatic cancer suitable for palliative antineoplastic therapy
* locally advanced/metastatic cancer with uncontrolled symptoms
* end-stage heart failure
* end-stage respiratory failure
* end-stage liver failure
* end-stage renal failure

Exclusion Criteria:

* not able to be administered the screening tool
* major psychiatric disorders
* informed consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of the Simplified Screening Tool (SST) with respect to the SIAARTI/NCCN screening tool (EST) | Through study completion, an average of 1 year
  BACKGROUND: The aims of this study were to evaluate the feasibility of an Emergency Department (ED)-initiated screening to identify seriously ill patients in need of palliative care (PC) and to develop a simplified screening tool (SST).
  METHODS: Eligible patients with a known diagnosis of chronic heart, lung, liver, and kidney failures, or advanced cancer, awaiting to be hospitalized after an ED visit, were assessed with both screening tools (ie, EST and SST).
  The outcome of this study is to evaluate the accuracy of the SST in identifying chronically ill patients in need of a palliative care assessment in the hospital setting.

SECONDARY OUTCOMES:
Accuracy of Surprise Question (SQ) | Through study completion, an average of 1 year
  BACKGROUND: The surprise question (SQ), "Would the investigator be surprised if this patient died within the next year?" is effective in identifying the end-stage disease patients and therefore potentially unmet palliative care needs. The SG is one of the criteria assessed by screening tools to identify people in need of palliative care assessment.
  METHODS: Eligible patients with a known diagnosis of chronic heart, lung, liver, and kidney failures, or advanced cancer, awaiting to be hospitalized after an ED visit, underwent an evaluation of life expectancy using the Surprise Question (SQ).
  The outcome of this study is to evaluate the accuracy of SQ in identifying palliative care patients in their last year of life.
Symptom control in palliative care patients | Through study completion, an average of 1 year
  BACKGROUND: Good symptom control is important for delivering effective palliative care METHODS: Patients with a diagnosis of chronic heart, lung, liver, and kidney failures, or advanced cancer, hospitalized after an ED visit, fully according to the screening tool score, in an acute palliative care unit due to uncontrolled symptoms
  OUTCOME MEASURE: Measurements will be aggregated to arrive at a comparison between admission and discharge times of:
  * frequency (n,%) of following symptoms: pain, activity, nausea, depression, anxiety, drowsiness, appetite, sense of well-being and shortness of breath
  * frequency (n,%) of use of pain killer, interventional procedures, palliative sedation
Intensity of symptoms in patients admitted in an acute palliative care unit | Through study completion, an average of 1 year
  BACKGROUND: Good symptom control is important for delivering effective palliative care METHODS: Patients with a diagnosis of chronic heart, lung, liver, and kidney failures, or advanced cancer, hospitalized after an ED visit, fully according to the screening tool score, in an acute palliative care unit due to uncontrolled symptoms OUTCOME MEASURE: Measurements will be aggregated to arrive at a comparison between admission and discharge times of the intensity of symptoms using the Edmonton Symptom Assessment System, that consists of nine verbal numerical scales (0 as minimum value/better outcome; 10 as maximum value/ worse outcome)
Survival of patients in need of palliative care assessment | Through study completion, an average of 1 year
  BACKGROUND: Acute palliative care units (APCU) are new programs aimed at improving palliative care in hospitalized patients. Although most deaths in palliative care patients with end-stage diseases are expected, no data are available on survival.
  METHODS: Eligible patients with a known diagnosis of chronic heart, lung, liver, and kidney failures, or advanced cancer, hospitalized after an ED visit, fully according to the screening tool score in an APCU, due to uncontrolled symptoms.
  OUTCOME MEASURE DESCRIPTION: The aim of this study is to evaluate the survival time (day, months, years) from APCU admission to death for any cause (overall survival).
Discharge and unplanned hospital readmissions of patients in need of palliative care assessment | Through study completion, an average of 1 year
  BACKGROUND: Discharge planning represents one of the most important and complex decisions for patients admitted to an acute palliative care unit (APCU).
  METHODS: Eligible patients with a known diagnosis of chronic heart, lung, liver, and kidney failures, or advanced cancer, hospitalized after an ED visit, fully according to the screening tool score, in an APCU.
  OUTCOME MEASURE DESCRIPTION:
  This study is to evaluate:
  * the frequency of discharge at home and to hospice care
  * the frequency of unplanned hospital readmissions of palliative care patients discharged from our APCU.
Clinical characteristics and outcomes of palliative care patients referred to an acute palliative care unit | Through study completion, an average of 1 year
  BACKGROUND: Acute palliative care units (APCU) admit patients for symptom control, the transition to palliative care programs (home or hospice care), or end-of-life care.
  METHODS: Patients with a known diagnosis of chronic heart, lung, liver, and kidney failures, or advanced cancer, hospitalized after an ED visit, fully according to the screening tool score, in an APCU.
  OUTCOME MEASURE: multiple measurements will be aggregated to arrive at one detailed description of:
  * frequency (n,%) of following symptoms: pain, activity, nausea, depression, anxiety, drowsiness, appetite, sense of well-being and shortness of breath
  * frequency (n,%) of discharge at home and to hospice care

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cotogni, MD, MSc, Principal Investigator — Pain Manage&Palliative Care Dept Anesthesia Molinette University Hospital Turin
Locations (1):
- Pain Management and Palliative Care, Department of Anesthesia, Intensive Care and Emergency, Molinette Hospital, University of Turin, Turin, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotogni P, DE Luca A, Evangelista A, Filippini C, Gili R, Scarmozzino A, Ciccone G, Brazzi L. A simplified screening tool to identify seriously ill patients in the Emergency Department for referral to a palliative care team. Minerva Anestesiol. 2017 May;83(5):474-484. doi: 10.23736/S0375-9393.16.11703-1. Epub 2017 Jan 17. PMID 28094484
- [Background] Au DH, Udris EM, Fihn SD, McDonell MB, Curtis JR. Differences in health care utilization at the end of life among patients with chronic obstructive pulmonary disease and patients with lung cancer. Arch Intern Med. 2006 Feb 13;166(3):326-31. doi: 10.1001/archinte.166.3.326. PMID 16476873
- [Background] Kahn JM, Benson NM, Appleby D, Carson SS, Iwashyna TJ. Long-term acute care hospital utilization after critical illness. JAMA. 2010 Jun 9;303(22):2253-9. doi: 10.1001/jama.2010.761. PMID 20530778
- [Background] Jassal SV, Watson D. Dialysis in late life: benefit or burden. Clin J Am Soc Nephrol. 2009 Dec;4(12):2008-12. doi: 10.2215/CJN.04610709. Epub 2009 Nov 5. PMID 19965545
- [Background] Glare PA, Chow K. Validation of a Simple Screening Tool for Identifying Unmet Palliative Care Needs in Patients With Cancer. J Oncol Pract. 2015 Jan;11(1):e81-6. doi: 10.1200/JOP.2014.001487. Epub 2014 Nov 12. PMID 25392521
- [Background] Cotogni P, De Luca A, Saini A, Brazzi L. Unplanned hospital admissions of palliative care patients: a great challenge for internal and emergency medicine physicians. Intern Emerg Med. 2017 Aug;12(5):569-571. doi: 10.1007/s11739-017-1671-3. Epub 2017 May 5. No abstract available. PMID 28477288